CLINICAL TRIAL: NCT03307564
Title: Evaluation of a Novel Absorbable Radiopaque Hydrogel in Patients Undergoing Image-guided Radiotherapy for Pancreatic Adenocarcinoma
Brief Title: Radiopaque Hydrogel in Patients Undergoing Radiotherapy for Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Augmenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J17144; IRB00151816 (Other: JHMIRB)
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: marking the interface between the pancreas and duodenum with TraceIT Tissue Marker in patients undergoing image-guided radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TraceIT tissue marker injection (Experimental): The TraceIT injection will be performed during the endoscopic fiducial placement which is the standard of care. CTs to serially confirm TraceIT positioning will be performed on the same day during patient visits for their middle (2nd or 3rd fraction) and last (5th fraction) radiation therapy treatments
  Interventions: Device: TraceIT tissue marker injection

INTERVENTIONS:
Device: TraceIT tissue marker injection — The TraceIT injection will be performed during the endoscopic fiducial placement which is the standard of care. CTs to serially confirm TraceIT positioning will be performed on the same day during patient visits for their middle (2nd or 3rd fraction) and last (5th fraction) radiation therapy treatments.

SUMMARY:
The goal of this pilot imaging study is to evaluate the visibility of marking the interface between the pancreas and duodenum with TraceIT Tissue Marker. Patients with a pathologically confirmed diagnosis of BR/LAPC (borderline resectable/locally advanced pancreatic cancer) pancreatic adenocarcinomas indicated for neo-adjuvant image-guided radiotherapy with SBRT (stereotactic body radiation therapy) will be enrolled. This study will thus set the stage for further investigations using the TraceIT Tissue Marker to avoid duodenum toxicity with imaging localization, enabling further dose intensification with SBRT or IMRT to improve the clinical outcomes in BR/LAPC.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma is now the third leading cause of cancer-related death, with a devastating 5-year overall survival (OS) rate of nearly 8%, despite having the 12th most common incidence of all malignancies in the United States. One-third of patients will present with borderline resectable or unresectable, locally advanced pancreatic cancer (BR/LAPC). In the cases of LAPC, chemotherapy with or without radiation may be recommended to improve the quality of life by relieving symptoms and extending survival. Despite aggressive combined modality therapy, the median survival remains between 9 and 15 months.

Current guidelines for the management of BR/LAPC patients include single- or multi-agent chemotherapy or chemoradiation (CRT) in sequence with chemotherapy. Results of studies comparing chemotherapy alone to CRT for patients with BR/LAPC are mixed. The importance of local control or delaying local progression on improving morbidity and possibly mortality in patients with pancreatic cancer is supported by autopsy data demonstrating that 30% of patients die of locally destructive disease. It follows that in the cases of LAPC, advanced radiation therapy techniques using dose-escalation with intensity modulated radiotherapy (IMRT) and stereotactic body radiotherapy (SBRT) are potential strategies to improve local control.

A consistent challenge to dose-escalation with IMRT (intensity modulation radiation therapy) or SBRT is the sensitivity of the surrounding gastrointestinal organs, particularly the small bowel which is directly adjacent to the head of the pancreas head of the pancreas (HOP). For BR/LAPC patients treated with CRT, advances in image guidance have provided the opportunity to safely deliver higher biologically effective doses of radiation therapy using IMRT of >70 Gy (57.25 Gy in 25 fractions, BED 70.36 Gy) compared to standard fractionation regimens (50.40 Gy in 28 fractions or 50 Gy in 25 fractions, BED 59.47 Gy and 60 Gy, respectively). Those patients who underwent dose-escalated CRT with BED>70 Gy, did have a superior OS compared to those receiving BED<70 Gy, supporting the utility of dose-escalation in improving long-term outcomes. SBRT involves a short course of radiation therapy, five fractions or less, and has demonstrated higher rates of local control compared to CRT in other disease sites. Early studies evaluating SBRT for pancreatic cancer utilized single fractions of 25 Gy, resulting in local control rates of 100% at 1 year but unacceptably high rates of gastrointestinal toxicity. More recently, hypofractionated SBRT (33 Gy total, 6.6 Gy daily fractions) has been evaluated and utilized by our group in an effort to reduce the toxicity of therapy, with results demonstrating nearly 80% rate of freedom from local progression at one year and an acceptable 11% long-term gastrointestinal toxicity. Outcomes with SBRT are thus promising; however, higher local control rates with dose-escalation may be achievable, but current practice is limited due to risks of toxicity.

The goal of this pilot imaging study is to evaluate the visibility of marking the interface between the pancreas and duodenum with TraceIT Tissue Marker. Patients with a pathologically confirmed diagnosis of BR/LAPC pancreatic adenocarcinomas indicated for neo-adjuvant image-guided radiotherapy with SBRT will be enrolled. This study will thus set the stage for further investigations using the TraceIT Tissue Marker to avoid duodenum toxicity with imaging localization, enabling further dose intensification with SBRT or IMRT to improve the clinical outcomes in BR/LAPC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. BR/LAPC pancreatic carcinoma disease
3. Radiotherapy or chemoradiotherapy for treatment of the disease is indicated with the intent for eventual surgical resection
4. Subjects Screening/Baseline laboratory testing must meet the following laboratory value criteria:

   1. White blood cell count: ≥ 3.0 x 109/L
   2. Absolute neutrophil count (ANC): ≥ 1.5 x 109/L
   3. Platelets: ≥ 100 x 109/L
   4. Total bilirubin: ≤ 2.0 times upper limit of normal (ULN)
   5. AST (Aspartate Aminotransferase) and ALT (Alanine Aminotransferase): ≤ 3.0 times institutional upper normal limit
   6. Serum creatinine: 1.5 times ULN (upper limit of normal)
   7. INR (international normalized ratio): < 1.5
   8. Serum pregnancy: Negative
   9. Hemoglobin: ≥ 8.0 g/dl
5. Zubrod Performance Status 0-2
6. Subject or authorized representative, has been informed of the nature of the study and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site.

Exclusion Criteria:

1. Previous thoracic radiotherapy
2. Any GI (gastrointestinal) abnormality that would interfere with the ability to access the injection site
3. Active gastroduodenal ulcer or watery diarrhea
4. Active bleeding disorder or a clinically significant coagulopathy defined as a PTT (Partial thromboplastin time) >35s or INR>1.4 or platelet count less than 100,000 per mm3.
5. Active inflammatory or infectious process involving the gastrointestinal tract based on positive diagnosis or suspected diagnosis in the presence of fever>38°C or WBC>12,000/uL.
6. Compromised immune system: WBC (white blood count) <4000/uL or >12,000/uL.
7. History of Chronic Renal Failure.
8. Documented history of uncontrolled diabetes (i.e., symptomatic hyperglycemia that cannot be medically managed, fasting blood glucose level above 300 mg/dL, and/or frequent swings between hyperglycemia and hypoglycemia)
9. Currently enrolled in another investigational drug or device trial that clinically interferes with this study.
10. Unable to comply with the study requirements or follow-up schedule.
11. Any condition or comorbidity that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the subject.
12. Pregnancy, breast-feeding, women of child-bearing age must use contraceptives

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, MD, Principal Investigator — Johns Hopkins SKCCC
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TraceIT Tissue Marker Injection
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TraceIT Tissue Marker Injection
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white/caucasian | 3
  asian | 1
  other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Where TraceIT Tissue Marker Placement Achieved
Description: Measured as number of patients where marking the interface between the pancreas and duodenum with TraceIT Tissue Marker in patients undergoing image-guided radiotherapy for BR/LAPC pancreatic adenocarcinoma was achieved.
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | TraceIT Tissue Marker Injection
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: immediate post-procedure period (approximately 3 hours after injection of hydrogel while patients in recovery/observation)
Arm/Group | TraceIT Tissue Marker Injection
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TraceIT Tissue Marker Injection (N=6)
nausea (Gastrointestinal disorders) | 1 (6) — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03307564/Prot_SAP_000.pdf